CLINICAL TRIAL: NCT02077140
Title: A Phase II, Dose-escalating, Randomized, Double-blind, Multicenter Study to Evaluate the Efficacy, Safety and Pharmacokinetic Profile of MDT-10013 Versus Standard of Care in the Treatment of Acute Postoperative Pain Following Bunionectomy
Brief Title: A Study of MDT-10013 in the Treatment of Acute Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P13-01
Record Dates: First submitted 2014-02-26; First posted 2014-03-04 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDT-10013 (Experimental): Subjects will receive MDT-10013.
  Interventions: Drug: MDT-10013
- Standard of Care (Active Comparator): Subjects will receive standard of care.
  Interventions: Drug: Standard of care for pain

INTERVENTIONS:
Drug: MDT-10013
  Arms: MDT-10013
Drug: Standard of care for pain
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MDT-10013 in men and women 18 to 80 years of age who are undergoing bunionectomy. The primary objective is to determine the analgesic efficacy of MDT-10013 compared with standard of care in the treatment of acute postoperative pain after subjects undergo bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged 18 to 80 years.
2. Has a body mass index from 18 kg/m2 to 40 kg/m2.
3. Is scheduled to undergo primary, unilateral, first metatarsal bunionectomy (osteotomy and internal fixation) with no additional collateral procedures.
4. Is classified by American Society of Anesthesiologists Physical Status Classification System as Class I or II.
5. Must meet the following criteria if female:

   * Is of non-childbearing potential, defined as any woman who has undergone surgical sterilization or is more than 2 years postmenopausal
   * If of childbearing potential, may be enrolled on the condition that results of a pregnancy test are negative at baseline (at Screening and before surgery) and that she is routinely using an effective method of birth control with a low failure rate (i.e., hormonal contraception, intrauterine device, condoms in combination with a spermicidal cream, or total sexual abstinence)
6. Has read, understood, and signed the informed consent prior to study entry.
7. Is mentally competent, reliable, and cooperative to undergo all visits and procedures scheduled in the study protocol and to record the required information.
8. Has medical history, physical examination, vital signs, laboratory tests, and 12-lead electrocardiograms (ECGs) that are normal or without clinically relevant abnormalities as per investigator's judgment.

Exclusion Criteria:

1. Is a female who is pregnant or breastfeeding.
2. Is not indicated for surgery because of an inflammatory process or risk of infection or delayed wound healing (e.g., autoimmune disorder).
3. Has a history of allergy or hypersensitivity to the components in the investigational product or to the opioid medication (oxycodone).
4. Before surgery, has current orthostatic hypotension (defined as systolic blood pressure decrease of at least 20 mm Hg or a diastolic blood pressure decrease of at least 10 mm Hg or an increase in heart rate by 20 beats per minute within 3 minutes of sitting up or standing).
5. Has severe asthma, defined as requiring frequent or ongoing treatment to control symptoms. Exercise-induced asthma or mild asthma not requiring ongoing treatment may not be exclusionary at the discretion of the investigator.
6. Has a current gastrointestinal disorder associated with bleeding, a history of such a disorder, or gastrointestinal inflammatory diseases as Crohn's disease or ulcerative colitis.
7. Has any clinically significant cardiovascular condition as evidenced by physical examination, medical history, and/or baseline ECG.
8. Has evidence of bradycardia as shown by heart rate of <50 beats per minute via screening ECG.
9. Has a known infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
10. Has a chronic pain condition that may interfere with the subject's assessment of pain postoperatively, as determined by the investigator.
11. Has any poorly controlled or serious medical conditions, psychiatric illnesses, or clinically significant laboratory values that, in the opinion of the investigator, could compromise the safety of the subject or the scientific integrity of the study (e.g., uncontrolled hypertension, autoimmune disease, or clinically relevant symptoms of thyroid dysfunction).
12. Has presence or history of local or systemic malignant disease in the past 5 years (history of basal cell carcinoma will be allowed).
13. Has impaired renal function (creatinine >1.5 times upper limit of normal).
14. Has chronic impairment liver function (aspartate aminotransferase or alanine aminotransferase >3 times upper limit of normal).
15. Has insulin-dependent diabetes or uncontrolled diabetes mellitus (glycosylated hemoglobin >7%).
16. Has leukopenia (<3500 leukocytes/μL).
17. Has current treatment with any of the following medications:

    1. Systemic corticosteroids (intranasal/inhaled steroids are acceptable).
    2. Immunosuppressant therapy to treat autoimmune diseases (e.g., rheumatoid arthritis, multiple sclerosis, myasthenia gravis, systemic lupus erythematosus, sarcoidosis, focal segmental glomerulosclerosis, Crohn's disease, Behcet's Disease, pemphigus, and ulcerative colitis).
    3. Oral or topical products that contain clonidine (e.g., Catapres).
    4. Herbal supplements that contain yohimbine.
    5. Anticoagulant/antiplatelet therapy (prophylactic aspirin at 81 mg/day is acceptable). If applicable, aspirin therapy should be held before and after the study procedure on the basis of the investigator's discretion.
    6. Antiepileptic drugs, antipsychotics, tricyclic antidepressants, monoamine oxidase inhibitors, lithium, and sulfonamides.
    7. Calcium channel blocker, digoxin, or beta-adrenergic blockers.
18. Has chronic use of opioids (including tramadol), defined as use 20 out of the last 30 days before study screening.
19. Has a history of or current diagnosis of epilepsy.
20. Has a known or suspected history of drug or alcohol abuse (as determined by the investigator).
21. Is judged by the investigator not to be a suitable candidate for study treatment and pain relief medication on the basis of medical history, concomitant medication, and concurrent systemic disease.
22. Is not stabilized on the following medications for at least 8 weeks prior to dosing: selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs).
23. Is unable to refrain from taking nonsteroidal anti inflammatory drugs (NSAIDs) or opioids within the 24-hour period prior to surgery.
24. Has participated in any other clinical trial in the 4 weeks prior to Screening.
25. Experiences any surgical complication that, in the opinion of the investigator, precludes implantation of MDT-10013.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Phoenix, Arizona
  - Research Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to enroll 3 sequential cohorts, the 4th cohort was added after data review from Cohort 1-3. In each cohort, 48 subjects were randomized in a 3:1 ratio (investigational vs. control). The investigational subjects were implanted MDT-10013 strips in surgical wound while control subjects received standard of care for pain control.
Groups:
- 1 MDT-10013 Strip (In Cohort 1): For the investigational subjects of Cohort 1, one MDT-10013 strip was sutured to the exterior of the capsule wall.
- 2 MDT-10013 Strips (In Cohort 2): For the investigational subjects of Cohort 2, one MDT-10013 strip was sutured to the exterior of the capsule and 1 strip was sutured to the interior capsule wall.
- 3 MDT-10013 Strips (In Cohort 3): For the investigational subjects of Cohort 3, one MDT-10013 strip was sutured to the exterior of the capsule and 2 strips were sutured to the interior capsule wall.
- 2 MDT-10013 Strips (In Cohort 4): For the investigational subjects of Cohort 4, two strips were sutured to the interior capsule wall.
- Control (In Cohort 1-4): Control subjects in Cohort 1 to 4 received standard of care (no strip) for pain control.
Period: Overall Study
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1-4)
Started | 36 | 36 | 36 | 36 | 48
Completed | 32 | 34 | 34 | 32 | 43
Not Completed | 4 | 2 | 2 | 4 | 5
Not completed — Lost to Follow-up | 4 | 1 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- 2 MDT-10013 Strips (In Cohort 4): For the investigational subjects of Cohort 4, two MDT-10013 strips were sutured to the interior capsule wall.
- Control (In Cohort 1 to 4): Control subjects in Cohort 1 to 4 received standard of care for pain control.
- Total: Total of all reporting groups
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4) | Total
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 48 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (13.22) | 39.7 (11.90) | 40.4 (12.37) | 41.1 (13.49) | 40.7 (11.78) | 41.8 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 29 | 31 | 43 | 168
  Male | 4 | 3 | 7 | 5 | 5 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American-Indian or Alaska Native | 0 | 2 | 2 | 0 | 0 | 4
  Asian | 0 | 2 | 1 | 0 | 0 | 3
  Black or African-American | 4 | 4 | 7 | 5 | 4 | 24
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  White | 31 | 28 | 26 | 30 | 44 | 159
  Other | 0 | 0 | 0 | 0 | 0 | 0
  Data missing | 1 | 0 | 0 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: lbs] | 72.71 (15.41) | 71.97 (12.79) | 73.94 (14.51) | 72.99 (13.30) | 76.12 (14.24) | 73.71 (14.02)
Height [Mean (Standard Deviation); unit: cm] | 162.8 (8.12) | 162.5 (7.38) | 163.8 (8.92) | 162.8 (9.86) | 165.2 (8.67) | 163.5 (8.61)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (4.82) | 27.3 (4.51) | 27.4 (4.07) | 27.6 (4.44) | 28.0 (4.55) | 27.6 (4.45)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Over 1- 48hrs (SPI-48) From Cohort 1 to 3
Description: Summed pain intensity is a time-weighted average pain score in numeric rating scale (NRS) over 1 to 48hrs (SPI-48). Summed pain intensity is calculated as area under the curve, using the trapezoidal rule to bridge adjacent time points. Specifically, NRS scores for two adjacent time points are averaged and then multiplied by the time span between points (in hours). The theoretical range for SPI-48 is 0 to 470, with lower scores indicative of less pain over this time period (i.e., lower scores are consistent with better analgesia). Time 0 was defined as the time the capsule was closed.
Time Frame: over 1 to 48hrs
Population: The primary efficacy analysis was based on the Full Analysis dataset of Cohort 1 to 3. Full Analysis dataset included Safety population (i.e., all subjects who received at least 1 MDT-10013 strip or completed surgery in a standard-of-care group based on the actual treatment a subject received) having at least 1 postoperative pain assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control (In Cohort 1-3): Control subjects in Cohort 1 to 3 received standard of care for pain control.
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1-3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
units on a scale | 252.29 (74.423) | 213.28 (73.330) | 191.97 (84.940) | 215.35 (66.133)

2. Primary Outcome: Summed Pain Intensity Over 1- 48hrs (SPI-48)--Sensitivity Analysis Using Last Observation Carried Forward (LOCF)
Description: Similar to SPI-48, the theoretical range for this LOCF adjustment for rescue medication is 0-470, with lower scores indicative of less pain over this time period (i.e., lower scores are consistent with better analgesia). The calculation is identical to SPI-48 in terms of area-under the curve using the trapezoidal rule. However, the NRS score at the final assessment prior to rescue is carried forward through 48 hours, replacing the raw NRS scores post-rescue for each patient as applicable.
Time Frame: over 1 to 48hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control (In Cohort 1 to 3): Control subjects in Cohort 1 to 3 received standard of care for pain control.
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
units on a scale | 324.82 (65.141) | 284.60 (80.080) | 281.03 (82.593) | 281.83 (91.415)

3. Primary Outcome: Integrated Summed Pain Intensity Over 1- 48hrs (SPI-48) and Total Opioid Intake in First 48hrs --Sensitivity Analysis Using Silverman Method
Description: This sensitivity analysis is an integrated assessment of summed pain intensity over 1 to 48hrs (SPI-48) and total opioid intake (ME0-48) in first 48hrs. Briefly, subjects were ranked according to SPI-48 regardless of the treatment received (including Standard of Care, SOC). The mean of all the ranks for this variable was calculated. Then, the percent difference for each individual rank from the pooled mean rank was computed. This process was repeated for total opioid intake in the first 48hrs (ME0-48). The integrated endpoint for each subject was the sum of the rank order percent differences for SPI-48 and ME0-48. The theoretical minimum and maximum on the integrated endpoint are -197% and +197% in this study. Lower scores are better, indicative of less pain and/or less opioid intake.
Time Frame: over 1 to 48hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
percent difference | 23.66 (54.274) | -4.79 (55.043) | -17.36 (62.466) | -1.51 (52.306)

4. Primary Outcome: Summed Pain Intensity Over 1- 48hrs (SPI-48)--Sensitivity Analysis Using Windowed Worst Observation Carried Forward (WOCF)
Description: Similar to SPI-48, the theoretical range for this WOCF adjustment for rescue medication is 0-470, with lower scores indicative of less pain over this time period (i.e., lower scores are consistent with better analgesia). The calculation is identical in terms of area-under the curve using the trapezoidal rule. However, the NRS score at the final assessment prior to each instance of rescue medication is carried forward through for a window based on the approximate half-life of the drug, replacing the raw NRS scores post-rescue for each patient until the end of the pharmacological activity window, at which point calculations revert to raw NRS as applicable. Note that WOCF SPI-48 may include multiple adjustment windows for each patient, depending on the number or rescue events and the active life of the medication selected.
Time Frame: over 1 to 48hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
units on a scale | 322.08 (93.298) | 278.44 (83.515) | 257.57 (100.430) | 302.54 (82.105)

5. Secondary Outcome: Summed Pain Intensity Scores Over 1- 24hrs (SPI-24), 1- 72hrs (SPI-72) and 1- 96hrs (SPI-96)
Description: The theoretical range for SPI-24, SPI-72, and SPI-96 is 0 to 230, 0-710, and 0-960, respectively, with lower scores indicative of less pain over this time period (i.e., lower scores are consistent with better analgesia). Summed pain intensity is calculated as area under the curve, using the trapezoidal rule to bridge adjacent time points. Specifically, NRS scores for two adjacent time points are averaged and then multiplied by the time span between points (in hours).
Time Frame: over 1 to 24hrs, 1 to 72hrs, and 1 to 96hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
units on a scale
  SPI-24 | 132.18 (35.321) | 110.83 (35.831) | 102.42 (38.324) | 118.13 (33.591)
  SPI-72 | 325.96 (113.416) | 285.50 (109.126) | 259.42 (126.691) | 282.90 (105.476)
  SPI-96 | 393.29 (155.314) | 345.50 (144.692) | 322.97 (168.672) | 344.90 (147.835)

6. Secondary Outcome: Total Use of Opioid Analgesia Over 0 to 24hrs, 0 to 48hrs, 0 to 72hrs, and 0 to 96hrs.
Description: Total use of opioid analgesia over 0 to 24hrs, 0 to 48hrs, 0 to 72hrs, and 0 to 96hrs. The analgesia administered was converted to a morphine equivalent by using a standard conversion table.
Time Frame: over 0 to 24hrs, 0 to 48hrs, 0 to 72hrs, and 0 to 96hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: morphine mg equivalent
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
morphine mg equivalent
  Total opioid analgesia use over 0 to 24 hrs | 51.04 (21.798) | 37.64 (21.654) | 34.17 (18.927) | 55.42 (19.987)
  Total opioid analgesia use over 0 to 48 hrs | 81.67 (38.526) | 59.10 (32.278) | 56.04 (34.040) | 82.08 (34.203)
  Total opioid analgesia use over 0 to 72 hrs | 95.35 (50.886) | 73.68 (45.773) | 69.58 (46.876) | 95.63 (45.862)
  Total opioid analgesia use over 0 to 96 hrs | 106.04 (57.744) | 81.98 (54.366) | 77.92 (54.803) | 102.92 (51.805)

7. Secondary Outcome: Time to First Use of Opioid Analgesia
Time Frame: up to 96hrs
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
hours | 4.4 [3.3 to 5.1] | 5.3 [4.5 to 6.3] | 5.1 [4.3 to 5.9] | 3.7 [3.2 to 4.3]

8. Secondary Outcome: Subject's Satisfaction With Study Treatment
Description: Subject's satisfaction with study treatment as measured by a 5-point categorical scale where 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent
Time Frame: up to 72hrs
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | Control (In Cohort 1 to 3)
Number analyzed (Participants) | 36 | 36 | 36 | 36
Participants
  Poor | 11 | 3 | 3 | 9
  Fair | 3 | 5 | 4 | 6
  Good | 10 | 9 | 11 | 10
  Very good | 8 | 11 | 13 | 8
  Excellent | 4 | 8 | 5 | 3

9. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-t)
Description: Blood samples were taken for pharmacokinetic parameters of MDT-10013 determinations before surgery on Day 0; at 1, 2, 4, 6, 8, 12, 24, 48, 72, and 96 hours after Time 0 (96-hour sample for Cohort 4 only); and on Days 7 to 10 after Time 0. Time 0 was defined as the time the capsule was closed. Actual sampling times after T0 (to 1/1000th of an hour) were used to calculate PK parameters.
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36
h*pg/mL | 73885.02 (16743.59) | 127987.04 (36290.88) | 174207.74 (45114.71) | 144138.55 (40723.92)

10. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-∞)
Description: as for outcome 9
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 30 | 21 | 18 | 35
h*pg/mL | 79553.78 (18857.19) | 130511.64 (27496.95) | 216167.36 (72319.99) | 166887.29 (47337.97)

11. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 9
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36
pg/mL | 620.98 (135.36) | 1057.91 (269.09) | 1492.96 (470.27) | 1304.46 (360.07)

12. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Time to Maximum Plasma Concentration Observed (Tmax)
Description: as for outcome 9
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Median (Full Range); unit: hrs
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36
hrs | 48.1 [12.1 to 72.2] | 48.1 [12.1 to 72.2] | 60.2 [12.2 to 72.5] | 48.2 [24.1 to 72.5]

13. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Lag Time Before First Measurable Drug Concentration (Tlag)
Description: as for outcome 9
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Median (Full Range); unit: hrs
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36
hrs | 1.07 [0.00 to 2.08] | 0.00 [0.00 to 1.15] | 0.00 [0.00 to 2.08] | 1.05 [0.00 to 2.08]

14. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Terminal Plasma Half-life (t½)
Description: Blood samples were taken for pharmacokinetic parameters of MDT-10013 determinations before surgery on Day 0; at 1, 2, 4, 6, 8, 12, 24, 48, 72, and 96 hours after Time 0 (96-hour sample for Cohort 4 only); and on Days 7 to 10 after Time 0. Time 0 was defined as the time the capsule was closed.
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 30 | 21 | 18 | 35
hrs | 49.03 (7.32) | 52.28 (7.10) | 61.67 (16.79) | 50.55 (6.34)

15. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of MDT-10013: Terminal Phase Rate Constant (λz)
Description: as for outcome 14
Time Frame: up to 10 days
Population: PK analysis population consisted of all subjects who had PK samples analyzed.
Measure: Mean (Standard Deviation); unit: /hr
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4)
Number analyzed (Participants) | 30 | 21 | 18 | 35
/hr | 0.0144 (0.0021) | 0.0135 (0.0019) | 0.0118 (0.0025) | 0.0139 (0.0017)

16. Other Pre Specified Outcome: Summed Pain Intensity Scores (Exploratory Analysis)
Description: The theoretical range for SPI-24, SPI-48, SPI-72, and SPI-96 is 0 to 230, 0-470, 0-710, and 0-960, respectively, with lower scores indicative of less pain over this time period (i.e., lower scores are consistent with better analgesia). Summed pain intensity is calculated as area under the curve, using the trapezoidal rule to bridge adjacent time points. Specifically, NRS scores for two adjacent time points are averaged and then multiplied by the time span between points (in hours).
Time Frame: over 1 to 24hr, 1 to 48 hrs, 1 to 72hrs, and 1 to 96hrs
Population: The efficacy analyses of Cohort 1 to 4 were considered for exploratory analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control (In Cohort 1 to 4): Control subjects of Cohort 1 to 4 received standard of care for pain control.
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 48
units on a scale
  SPI-24 | 132.18 (35.321) | 110.83 (35.831) | 102.42 (38.324) | 98.39 (33.481) | 116.94 (37.117)
  SPI-48 | 252.29 (74.423) | 213.28 (73.330) | 191.97 (84.940) | 205.83 (72.126) | 218.35 (74.235)
  SPI-72 | 325.96 (113.416) | 285.50 (109.126) | 259.42 (126.691) | 291.17 (113.586) | 290.44 (116.649)
  SPI-96 | 393.29 (155.314) | 345.50 (144.692) | 322.97 (168.672) | 369.17 (157.870) | 354.60 (161.791)

17. Other Pre Specified Outcome: Total Use of Opioid Analgesia (Exploratory Analysis).
Time Frame: over 0 to 24hrs, 0 to 48hrs, 0 to 72hrs, and 0 to 96hrs
Population: The efficacy analyses of Cohort 1 to 4 were considered for exploratory analyses.
Measure: Mean (Standard Deviation); unit: morphine mg equivalent
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 48
morphine mg equivalent
  Total opioid analgesia use over 0 to 24 hrs | 51.04 (21.798) | 37.64 (21.654) | 34.17 (18.927) | 40.00 (19.558) | 52.66 (20.082)
  Total opioid analgesia use over 0 to 48 hrs | 81.67 (38.526) | 59.10 (32.278) | 56.04 (34.040) | 65.63 (33.845) | 76.41 (33.314)
  Total opioid analgesia use over 0 to 72 hrs | 95.35 (50.886) | 73.68 (45.773) | 69.58 (46.876) | 85.56 (50.611) | 90.16 (44.586)
  Total opioid analgesia use over 0 to 96 hrs | 106.04 (57.744) | 81.98 (54.366) | 77.92 (54.803) | 103.47 (67.189) | 97.34 (50.863)

18. Other Pre Specified Outcome: Time to First Use of Opioid Analgesia (Exploratory Analysis)
Time Frame: up to 96hrs
Population: The efficacy analyses of Cohort 1 to 4 were considered for exploratory analyses.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 48
hours | 4.4 [3.3 to 5.1] | 5.3 [4.5 to 6.3] | 5.1 [4.3 to 5.9] | 5.1 [3.7 to 5.9] | 4.2 [3.2 to 4.4]

19. Other Pre Specified Outcome: Subject's Satisfaction With Study Treatment (Exploratory Analysis)
Description: as for outcome 8
Time Frame: up to 72hrs
Population: The efficacy analyses of Cohort 1 to 4 were considered for exploratory analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4)
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 48
Participants
  Poor | 11 | 3 | 3 | 8 | 10
  Fair | 3 | 5 | 4 | 4 | 7
  Good | 10 | 9 | 11 | 8 | 17
  Very good | 8 | 11 | 13 | 10 | 10
  Excellent | 4 | 8 | 5 | 6 | 4

ADVERSE EVENTS:
Time Frame: up to 3 months
Groups:
- Control (In Cohort 1 to 4): Control subjects in Cohort 1 to 4 received standard of care (no strip) for pain control.
Arm/Group | 1 MDT-10013 Strip (In Cohort 1) | 2 MDT-10013 Strips (In Cohort 2) | 3 MDT-10013 Strips (In Cohort 3) | 2 MDT-10013 Strips (In Cohort 4) | Control (In Cohort 1 to 4)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/48
Other Adverse Events (participants affected / at risk) | 28/36 | 34/36 | 30/36 | 24/36 | 38/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 MDT-10013 Strip (In Cohort 1) (N=36) | 2 MDT-10013 Strips (In Cohort 2) (N=36) | 3 MDT-10013 Strips (In Cohort 3) (N=36) | 2 MDT-10013 Strips (In Cohort 4) (N=36) | Control (In Cohort 1 to 4) (N=48)
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 5 | 2 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 11 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 18 | 21 | 17 | 8 | 31
Paraesthesia oral (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 11 | 7 | 7 | 8
Chills (General disorders) | 0 | 1 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 1
Granuloma (General disorders) | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion site bruising (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal dryness (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 2 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 12 | 15 | 6 | 14
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 5 | 9 | 4 | 2 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 3 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 4 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 5
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 8
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 4
Hypotension (Vascular disorders) | 0 | 11 | 7 | 5 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less